CLINICAL TRIAL: NCT01795170
Title: Neurodevelopmental Outcome of Early Dietary Lysine Restriction in Pyridoxine
Brief Title: Neurodevelopmental Outcome of Early Dietary Lysine Restriction in Pyridoxine Dependent Epilepsy Patients
Acronym: NOEL
Status: Withdrawn | Type: Observational
Why Stopped: The study couldn't be initiated as we did not secure funding.
Sponsor: University of British Columbia (Other)
Collaborators: March of Dimes (Other); British Columbia Childrens Hospital Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: H12-03481
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Pyridoxine Dependant Epilepsy
Keywords: Pyridoxine Dependant Epilepsy; Antiquitin Deficiency; Lysine Restricted Diet
MeSH Terms: conditions — Pyridoxine-dependent epilepsy | interventions — Pyridoxine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test Group: Patients receiving a lysine restricted diet adjunct to pyridoxine therapy will be considered as participants in the 'exposure'/test group
  Interventions: Dietary Supplement: Lysine Restricted Diet; Drug: Pyridoxine
- Control Group: Patients on pyridoxine mono-therapy will be participants in the 'control' group
  Interventions: Drug: Pyridoxine

INTERVENTIONS:
Dietary Supplement: Lysine Restricted Diet — Daily lysine intake will be managed to maintain a plasma lysine level of 50-80 µmol/L (normal range: 52-196 µmol/L). Diet prescriptions will be based on international guidelines for glutaricaciduria type I, another inborn error of lysine catabolism. In order to meet the recommended daily protein intake (DRI) [23,24], the diet may include commercially available lysine-free amino acid formulas approved for use in conditions affecting lysine metabolism, as well as commercially available low-protein products based on the participant's taste.
  Groups: Test Group
Drug: Pyridoxine — All participants will be on 15-30 mg/kg/day of pyridoxine therapy up to a maximum of 500mg/day divided in 2-3 doses enterally

SUMMARY:
Restricting dietary lysine intake in infants from age 3 months or less with confirmed diagnosis of pyridoxine-dependent epilepsy due to Antiquitin (ATQ) deficiency will: reduce the accumulation of neurotoxic substratesα-aminoadipicsemialdehydeandits cyclic equivalent 1-piperideine-6-carboxylate;and will improve overall neurodevelopmental outcome at 3 years of age by acting as an effective intervention into the complex pathophysiology of the condition.

DETAILED DESCRIPTION:
I Purpose: The purpose of this multi-centre study is to further assess the safety and efficacy of the proposed lysine restricted diet in confirmed ATQ deficient PDE patients.

II Hypothesis: Restricting dietary lysine intake in infants from age 3 months or less with confirmed diagnosis of pyridoxine-dependent epilepsy due to Antiquitin (ATQ) deficiency will: reduce the accumulation of neurotoxic substratesα-aminoadipicsemialdehydeandits cyclic equivalent 1-piperideine-6-carboxylate;and will improve overall neurodevelopmental outcome at 3 years of age by acting as an effective intervention into the complex pathophysiology of the condition.

III Justification: We hope that participants have a much improved chance to avoid the same degree of developmental delay and associated problems. If this study demonstrates a significant improvement of normal development and proves to be safe to use this would provide a positive benefit to the child, the families involved as well as decreasing the burden on the health care system which currently must provide for life long care of these affected children.

IV Objectives: To determine the safety and efficacy of the lysine restricted diet on numerous primary and secondary outcome measures as listed in the protocol. The primary objective of this study is to evaluate neurodevelopmental outcome based on neuropsychological assessments using Bayley-III.

V Research Method:

1. Recruitement - Infants and/or children ranging from less than 3 months up to 3 years of age who have been diagnosed with PDE and with confirmed ATQ deficiency will be recruited within the 3 participating TIDE clinics (Medical Genetics, Biochemical Diseases, Neurology). Families may choose to participate in the TEST group or CONTROL group if they do not wish to undergo the lysine restricted diet regimen or decline to participate altogether.
2. Study visits - For participants in the TEST group, this will include a baseline visit and follow up visits at ages 3 months, 6 months then every 6 months until 3 years of age. For participants in the CONTROL group study visits include a baseline visit and 1 follow up visit at age 3 years. Routine clinical care visits can be scheduled as per treating physician's discretion at shorter intervals if needed.
3. Procedures: The following safety and efficacy measures will be performed at the specified study visits (Refer to table1 protocol or consent): medical history, vital signs, anthropometric measurements, Physical and Neurological exams, vision & hearing assessments, blood and urine samples tested for biomarkers, electroencephalogram, cognitive function test, ages and stages questionnaire, quality of life questionnaire, MRI, Cerebral Spinal fluid request only if lumbar puncture is being performed for clinical purposes.
4. Study Outcomes: The following outcomes will be measured.

Efficacy:

Primary Outcomes

* Neurocognitive development at age 3 years defined by total developmental index measured using the Bayley Scales for Infant and Toddler Development, 3rd Edition (Bayley-III)
* Level of biochemical marker-α- aminoadipic semialdehyde (AASA) its cyclic equivalent P6C in plasma and urine Secondary Outcomes
* Seizure frequency: clinical and electrical (EEG)
* Quality of life through a HR-QOL questionnaire
* Neurological deficits through neuro exam

Safety:

Primary Outcomes

* Anthropometric measures
* Plasma lysine and branched chain amino acid levels Secondary Outcomes
* Global nutritional assessment with plasma levels for albumin, prealbumin, total protein, iron parameters, zinc, selenium, CBC, folic acid, vitamin B12
* Peripheral sensory neuropathy (relevant because the lysine restriction is expected to reduce chemical inactivation of pyridoxine, thus potentially increasing the risk of toxicity)

VI Statistical Analysis:

I. OVERALL STUDY DESIGN Structure: We will conduct a multicenter, open label, negative-controlled observational cohort study to assess the safety and the efficacy on neurodevelopmental outcome of early dietary lysine restriction as an adjunct to pyridoxine therapy for infants with pyridoxine-dependent epilepsy resulting from ATQ deficiency.

Treatment Exposure: Patients receiving a lysine restricted diet adjunct to pyridoxine therapy will be considered as participants in the 'exposure'/test group and patients on pyridoxine mono-therapy will be participants in the 'control' group. The ratio of test participants to controls in the study will be 1:2.

Duration: All participants will be monitored for safety and neurodevelopmental outcome until the age of 3 years.

Efficacy & Safety Analysis: Data will be summarized with descriptive statistics, frequency tabulations, and data listings. Analyses include comparison of treatment effect before and after diet restriction within each participant, and comparison between test and control groups. Analysis will be performed on intent-to-treat population including all enrolled participants. The primary objective of this study is to evaluate neurodevelopmental outcome based on neuropsychological assessments using Bayley-III. The evaluation comprises the following scales: Cognitive Scale, Language Composite Scale with Receptive and Expressive Language subscales, and Motor Composite Scale with Fine- and Gross-Motor subscales. A composite score of all the scales gives the total developmental index. For the composite score and each scale, a hypothesis test can be performed to compare test group and the control group. A 2-sided 95% confidence interval for the mean change in Treatment minus mean change in control groups will be calculated for the total developmental index and each individual scale of Bayley-III to evaluate any particular nonnegative quantity of clinical interest. Similar analysis using appropriate parametric (ANOVA, ANCOVA, Fishers exact test) and nonparametric tests (Wilcoxon rank sum test) will be done for all efficacy and safety outcomes. Severity and relationship to treatment of the adverse events will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pyridoxine-dependent epilepsy based on clinical symptoms and elevated levels of plasma or urine AASA. Confirmation by at least one known disease causing mutation in the ALDH7A1 gene to be obtained within one month of enrollment.
* Participant is male or female <3 years of age.

  * Participants in the test arm have to be less than 3 months of age when the dietary restriction was started.
  * Participants in the control arm may be older than 3 months of age but must not be older than 3 years of age when they are enrolled into the study and must have been on pyridoxine treatment prior to age 3 months and not treated with dietary lysine restriction at any time during their life.
* Participant is managed with a vitamin B6 dose of 15-30 mg/kg/day continuously beginning at < 3 months age, and willing to maintain this dose for the study duration.
* Participants must have been offered dietary lysine restriction as adjunct therapy as part of standard clinical care.
* Parent(s) or guardian(s) is willing and able to provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures.

Exclusion Criteria:

* Diagnosis is not confirmed: Participant does not have a mutation in the ALDH7A1 gene.
* Participant was treated prenatally for PDE with pyridoxine (i.e. mother was on pyridoxine)
* Timing of dietary restriction: Participant is on a lysine-restricted diet from an age > 3months.
* Confounding factors:

  * Participant is a pre-term with a gestational age < 32 weeks
  * The participant has a birth weight less than the 2nd percentile or weighs less than 2nd percentile at study entrance (on age appropriate growth chart).
  * Participant shows an intracranial malformation or abnormality unrelated to ATQ deficiency, as diagnosed on the cranial ultrasound and/or MRI brain scan
  * Participant has any other disorder identified that can affect the cognitive function in the opinion of the coordinating principal investigators.
* A known allergy or sensitivity to any component of the products commonly used in a lysine-restricted diet or to other products associated with lysine restriction or any other products associated with general study procedures.
* Participant is on oral folinic acid and/or pyridoxal phosphate treatment at study entrance.
* Participant has any condition or situation which, in the investigator's opinion, places the patient at significant risk of adverse events, or may interfere significantly with their participation and compliance in the study.

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with pyridoxine-dependent epilepsy resulting from ATQ deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive development at age 3 years | 3 years
  defined by total developmental index measured using the Bayley Scales for Infant and Toddler Development, 3rd Edition (Bayley-III)
Level of biochemical marker-α- aminoadipicsemialdehyde (AASA) in plasma and urine | 3 years

SECONDARY OUTCOMES:
Seizure frequency: clinical and electrical (EEG) | 3 years
Quality of life | 3 years
Neurological deficits | 3 years

OTHER OUTCOMES:
Anthropometric measures | 3 years
Plasma lysine and branched chain amino acid levels | 3 years
Global nutritional assessment with plasma levels for albumin, prealbumin, total protein, iron parameters, zinc, selenium, CBC, folic acid, vitamin B12 | 3 years
Peripheral sensory neuropathy (relevant because the lysine restriction is expected to reduce chemical inactivation of pyridoxine, thus potentially increasing the risk of toxicity) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clara van Karnebeek, Principal Investigator — University of British Columbia; Sylvia Stockler, Principal Investigator — University of British Columbia
Locations (7):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Seattle Children's Hospital, Seattle, Washington
- BC Children's Hospital, Vancouver, British Columbia, Canada
- Hannover Medical School, Hanover, Hannover, Germany
- Maxima Medical Center, Veldhoven, Netherlands
- Kinderspital Zürich, Zurich, Switzerland
- University College London, London, United Kingdom

REFERENCES:
- [Background] van Karnebeek CD, Hartmann H, Jaggumantri S, Bok LA, Cheng B, Connolly M, Coughlin CR 2nd, Das AM, Gospe SM Jr, Jakobs C, van der Lee JH, Mercimek-Mahmutoglu S, Meyer U, Struys E, Sinclair G, Van Hove J, Collet JP, Plecko BR, Stockler S. Lysine restricted diet for pyridoxine-dependent epilepsy: first evidence and future trials. Mol Genet Metab. 2012 Nov;107(3):335-44. doi: 10.1016/j.ymgme.2012.09.006. Epub 2012 Sep 10. PMID 23022070